CLINICAL TRIAL: NCT01292421
Title: Pilot Study Testing the Immunogenic Efficacy of an Edible Vaccine for Hepatitis B in Healthy Volunteers
Brief Title: Edible Hepatitis B Vaccine Therapy in Healthy Participants Who Have Undergone Previous Vaccination
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: I 124207; NCI-2011-00064 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Hepatitis B Surface Antigens; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Placebo Comparator): Participants consume placebo HBV-EPV on days 0, 14, 28, and 56.
  Interventions: Other: placebo; Other: immunoenzyme technique
- Arm II (Experimental): Participants consume HBV-EPV expressing HBsAg on days 0 and 28 and placebo HBV-EPV on days 14 and 56.
  Interventions: Biological: hepatitis B antigen peptide; Other: placebo; Other: immunoenzyme technique
- Arm III (Experimental): Participants consume HBV-EPV expressing HBsAg on days 0, 28, and 56 and placebo HBV-EPV on day 14.
  Interventions: Biological: hepatitis B antigen peptide; Other: placebo; Other: immunoenzyme technique
- Arm IV (Experimental): Participants consume HBV-EPV expressing HBsAg on days 0, 14, 28, and 56.
  Interventions: Biological: hepatitis B antigen peptide; Other: immunoenzyme technique

INTERVENTIONS:
Biological: hepatitis B antigen peptide — Given PO
  Other Names: HBsAg; peptide, hepatitis B antigen
  Arms: Arm II; Arm III; Arm IV
Other: placebo — Given orally (PO)
  Other Names: PLCB
  Arms: Arm I; Arm II; Arm III
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques

SUMMARY:
RATIONALE: Hepatitis B antigen peptide (HBsAg) vaccine may help the body build an immune response and help prevent hepatitis B. PURPOSE: This clinical trial studies edible HBsAg vaccine therapy in healthy participants who have undergone previous vaccination.

DETAILED DESCRIPTION:
OBJECTIVES: I. To evaluate the safety, tolerability, and immunogenicity of orally delivered HBsAg that is formulated as an expressed protein in transgenic potato tubers (HBV-EPV) at different doses and schedules. OUTLINE: Patients are randomized to 1 of 4 treatment arms. ARM I: Participants consume placebo HBV-EPV on days 0, 14, 28, and 56. ARM II: Participants consume HBV-EPV expressing HBsAg on days 0 and 28 and placebo HBV-EPV on days 14 and 56. ARM III: Participants consume HBV-EPV expressing HBsAg on days 0, 28, and 56 and placebo HBV-EPV on day 14. ARM IV: Participants consume HBV-EPV expressing HBsAg on days 0, 14, 28, and 56. After completion of study treatment, patients are followed up at days 70, 84, 98, and 114.

ELIGIBILITY:
Inclusion Criteria:

* All Roswell Park Cancer Institute (RPCI) staff, faculty, and students, who are in good health
* Participants confirmation of history of primary immunization series with recombinant hepatitis B (HB) vaccine (last dose at least one year prior to screening anti-HBs level assessment)
* Current anti-HBs levels less than or equal to 115 mIU/mL
* Major organ functions within acceptable medical limits as determined in routine clinical laboratory screening tests
* Expected availability for the duration of the study period
* If female, then documentation that the subject is not pregnant by an acceptable laboratory test and that the subject is using an adequate birth control method to prevent pregnancy for at least 3 months following the last immunization in the study
* Human immunodeficiency virus (HIV) antibody negative
* Ability to provide written informed consent
* Supervisor approval

Exclusion Criteria:

* Known history of allergy or hypersensitivity to potato, potato components or potato products
* Known history of allergy to hepatitis B vaccine in any form or to components of hepatitis B vaccine
* Pregnancy or breast feeding
* Current anti-HBS levels greater than 115 mIU/mL
* Known immunodeficiency, cancer, or use of immunosuppressive medication including cancer chemotherapy and systemic steroids (excluding intermittent use of topical steroids)
* Participation in another investigational study within 30 days of enrollment in this study
* Known and currently active gastrointestinal disease including any of the following: peptic ulcer disease, gastroesophageal reflux, inflammatory bowel disease, diverticulitis, or pancreatitis
* Use of prescription medication or over the counter H2 blockers or proton pump inhibitors (PPIs) for any of the above diseases regularly and within 1 month of enrollment
* Diagnosis of insulin-dependent diabetes or multiple sclerosis
* Significant laboratory abnormality which suggests dysfunction of hematological, renal, or hepatic systems
* Known history of hepatitis B infection in the past
* Temporary exclusion for mild upper respiratory illness, gastrointestinal illness, or other febrile episode that is expected and documented to resolve

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Maximum fold increase in anti-HBsAg titer levels relative to baseline levels | Over 70 days

SECONDARY OUTCOMES:
Absolute maximum response | On days 0, 7, 14, 21, 28, 35, 42, 56 70, 84, 98, and 114
Area under the curve | On days 0, 7, 14, 21, 28, 35, 42, 56 70, 84, 98, and 114
Proportion of two-fold responses in anti-HBsAg titer levels | On days 0, 7, 14, 21, 28, 35, 42, 56 70, 84, 98, and 114

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, Principal Investigator — Roswell Park Cancer Institute